CLINICAL TRIAL: NCT07018349
Title: Low Dose Oral Minoxdil in Androgenic Alopecia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Hala Batool, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.F.2-81/2025-GENL/258/JPMC
Record Dates: First submitted 2025-06-01; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Androgenetic Alopecia (AGA)
Keywords: androgenetic alopecia (AGA); Minoxdil; Low oral doses
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Intervention Model Description: AGA patients will be randomly allocated in both groups using the envelopes method to reduce the biasness. For 3-months, patients in Group-A will get 2.5mg of minoxidil once daily, while those in Group-B will receive 1mg of minoxidil once daily orally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Minoxidil 2.5% mg (Experimental): Group-A: 2.5% mg of minoxidil once daily, orally.
  Interventions: Drug: 2.5% Oral minoxidil
- Oral Minoxidil 1% mg (Experimental): Group-B: 1% mg of minoxidil once daily orally.
  Interventions: Drug: 1% Oral Minoxidil

INTERVENTIONS:
Drug: 2.5% Oral minoxidil — AGA patients will be randomly allocated in both groups using the envelopes method to reduce the biasness. For 3-months, patients in Group-A will get 2.5mg of minoxidil once daily, while those in Group-B will receive 1mg of minoxidil once daily orally. After starting therapy, patients will be asked to come back for evaluations 3 months later. Safety, satisfaction, and the effects of the treatment will be reported. Final outcomes will be evaluated at 3 months post treatment.
  Arms: Oral Minoxidil 2.5% mg
Drug: 1% Oral Minoxidil — Group-B will receive 1mg of minoxidil once daily orally
  Arms: Oral Minoxidil 1% mg

SUMMARY:
In order to successfully treat androgenetic alopecia (AGA), this study compares the efficacy of low-dose oral minoxidil dosages of 0.25 mg and 1 mg. It addresses a critical gap in current research, as few studies have examined the relationship between low dosage and outcomes like hair diameter, density, patient satisfaction, and adverse effects, including hypertrichosis. Previous research suggests that low dose of oral minoxidil is a safe and well-tolerated option for hair loss, but the optimal dose for maximizing benefits while minimizing side effects remains unclear. This study aims to determine which dose offers the best balance of efficacy and safety for AGA patients.

DETAILED DESCRIPTION:
The most prevalent kind of progressive hair loss, androgenetic alopecia (AGA), is becoming more prevalent with growing age. AGA can affect a person's quality of life. For men, it shows up as a noticeable receding frontal hairline, whereas for women, it shows up as overall hair loss with frontal hairline retention. The primary causes of the condition are 5-alpha-reductase and dihydrotestosterone (DHT), which shorten anagen cycles and decrease hair follicles. It is still unclear whether precise processes underlie AGA start and vulnerability. AGA is thought to be a polygenic disorder whose onset and progression are influenced by the interplay of environmental, endocrine, and genetic variables. Several studies have shown that AGA negatively impacts on the quality of life (QoL) and self-esteem of the patients. However, because patients' expectations of treatment outcomes are typically higher than reality, AGA has continued to be a therapeutic problem for dermatologists.

FDA-approved treatment managements for AGA at present include oral finasteride, topical minoxidil 2%-5%, and low-level light therapy. The most often recommended drug among them is topical minoxidil solution. The selection of treatments for androgenetic alopecia therapy is still difficult as it requires moral, evidence-based judgment and takes into account the demands, compliance, financial constraints, degree of hair loss, and cosmetic preferences of each patient. Despite the fact that there are several medication, surgery, light-based, and nutraceutical treatment options available to stop or reverse the progression of AGA, selecting the best treatments for this chronic condition can be challenging. This study aims to determine which dose offers the best balance of efficacy and safety for AGA patients.

This study will be an RCT study. All patients will be adequately informed about the treatment regimen, follow-ups, and likely adverse effects before the start of the study. A written consent form will be obtained from each patient.

The study's eligibility for participation will be assessed for patients with AGA with the severity ranging from mild to moderate AGA. All AGA patients will get a trichoscopy and a complete scalp examination on their first appointment in order to rule out other hair-loss conditions, such as other types of alopecia like scarring or inflammatory and alopecia areata. Each patient's AGA stage will then be ascertained using the Savin scale for female patients and the "Norwood Hamilton scale" for male patients. Individuals who meet the clinical and trichoscopic criteria for mild to moderate AGA will be assessed for trial eligibility. Before beginning therapy, testing for hematological disorders, liver, kidney, thyroid, electrolytes, and pregnancy will be conducted. At 3-month follow-up appointment, measurements of body weight and blood pressure will also be taken.

AGA patients will be randomly allocated in both groups using the envelopes method to reduce the biasness. For 3-months, patients in Group-A will get 2.5mg of minoxidil once daily, while those in Group-B will receive 1mg of minoxidil once daily orally. After starting therapy, patients will be asked to come back for evaluations 3 months later. Safety, satisfaction, and the effects of the treatment will be reported. Final outcomes will be evaluated at 3 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a clinical and trichoscopic diagnosis of mild to severe AGA

Exclusion Criteria:

* Patients who, within three months before the trial, had undergone systemic or topical therapies for AGA
* People who suffer from additional hair loss conditions such hyperandrogenism, scarring or inflammatory alopecia, or any hormonal disorders.
* Sensitivity to minoxidil
* Patients with history of severe systemic diseases (heart, renal, or hepatic), a history of hypertension or hypotension, pregnant and breast-feeding women will also be excluded.
* Patient who will not be willing to provide written informed consents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Hair count and Thickness | 3 months
  Three distinct areas of the scalp will be marked with jet black Micropigment to guarantee precise measurements. These sites, which will be called the vertex points, mid-frontal, and frontal, respectively, were situated 12, 16, and 24 cm from the glabella. Following the application of just one drop of pigment to the selected area, the ink will be tattooed onto the skin using an insulin needle. The tattooed regions were photographed from a distance using a dermoscopic gadget (FotoFinder System Gmbh) that was linked to a camera (Canon EOS M100 DSLR) and a mobile phone. A trichology-trained technician who was blind to the process manually counted the number of hairs in a 1 cm 2 area surrounding each marked spot. Five randomly chosen hairs near the tattooed region will have their thicknesses measured with 3D-Slicer software, and the results will be averaged.
Photographic assessment | 3 month
  A standardized global pretreatment picture of the mid-anterior scalp will be taken using a digital camera in a fixed position, with the use of stereotactic positioning equipment, illumination, and styling. Additionally, close-up pictures of the tattooed areas will be taken at 12cm, 16cm, and 24cm from the glabella. A standardized seven-point rating system was used by two blind investigators to evaluate the photos separately.

SECONDARY OUTCOMES:
Patient satisfaction | 3 month
  On a scale of 1 to 10, where 10 denotes the highest level of satisfaction and 1 denotes the lowest, patients will be assessed how satisfied they are with the effects of their treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinnah PMC, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No